CLINICAL TRIAL: NCT01798160
Title: Selective Internal Radiation Therapy (SIRT) Versus Transarterial Chemoembolisation (TACE) for the Treatment of Hepatocellular Carcinoma (HCC).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Michael Bernhard Pitton, Consultant, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRT-TACE-HCC-Mainz-1
Record Dates: First submitted 2013-02-16; First posted 2013-02-25 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic; Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB TACE (Active Comparator): Drug eluting Beads (DC Beads) loaded with Doxorubicin
  Interventions: Procedure: DEB TACE
- SIRT (Experimental): Selective Internal Radiation Therapy using Yttrium 90 loaded resin beads (Sir Spheres)
  Interventions: Procedure: SIRT

INTERVENTIONS:
Procedure: DEB TACE — DEB TACE every 6 weeks until either no viable tumor or endpoint reached.
  Other Names: Chemoembolization
  Arms: DEB TACE
Procedure: SIRT — Selective Internal Radiation Therapy once at the beginning of the study. Follow up until endpoint.
  Other Names: Radioembolization
  Arms: SIRT

SUMMARY:
Selective Internal Radiation Therapy is superior to Transarterial Chemoembolisation for the treatment of intermediate stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* HCC, proven by histology or according to EASL criteria
* Intermediate stage HCC (stage B according to BCLC)
* At least one measurable lesion in magnetic resonance imaging (MRI)
* Tumor load ≤ 50%
* preserved liver function (Child Pugh A and B)

Exclusion Criteria:

* Patients feasible for curative treatment (e.g. resection or local ablation)
* Previous TACE or SIRT
* Chemotherapy during the last 4 weeks
* Child Pugh stage C
* BCLC stage D
* ECOG Performance Status >0
* Tumor involvement >50% of the liver
* Extrahepatic tumor
* Serum Bilirubin >2.0 mg/dl; Serum Albumin 2.8 g/dl, Serum Creatinine >2 mg/dl; Leukocytes <3000/ml; Thrombocytes <50000/ml
* Clinically apparent ascites (ascites only in CT/MRI is no exclusion criteria)
* Esophageal bleeding during the last 3 months
* Hepatic encephalopathy
* Transjugular intrahepatic portosystemic shunt (TIPS)
* Infiltration or occlusion of the portal vein
* Hepatofugal blood flow in the portal vein
* Hepatopulmonary shunt ≥ 20% in the macroaggregated albumin scan
* Contraindications against angiography
* Gravidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Progression-free-Survival | up to three years
Overall-Survival | up to three years